CLINICAL TRIAL: NCT00175799
Title: Validation of Severity of Illness Scoring Systems in Paediatric Intensive Care Units in Canada Outcome: Validation and Comparison of 2 Severity of Illness Scores in Canadian PICU Population
Brief Title: Validation of Severity of Illness Scoring Systems in Paediatric Intensive Care Units in Canada
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H03-70601; 04-1310
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Intensive Care Units, Pediatric
Keywords: Observational study of physiological status at entry into PICU as a predictor of outcome, comparison of two commonly used scores (PRISM and PIM); Data from children admitted to a Paediatric Intensive Care unit

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of the validation of severity of illness scoring systems in Paediatric Intensive Care Units (PICUs) in Canada.

DETAILED DESCRIPTION:
Outcome: Validation and comparison of 2 severity of illness scores in a Canadian PICU population.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to participating PICUs over a 1 year period.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children admitted to participating PICUs over a 1 year period.
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wensley, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital ICU Dept., Vancouver, British Columbia, Canada